CLINICAL TRIAL: NCT00729339
Title: Role of Mosapride in Patients With Gastroesophageal Reflux Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lotung Poh-Ai Hospital (Other)
Collaborators: Tomorrow Medical Foundation (Other)
Responsible Party: Hsin-Hong Chen/Superintendent, Lotung Poh-Ai Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: OMCP-97-011
Record Dates: First submitted 2008-07-31; First posted 2008-08-07 (Estimated); Last update posted 2009-05-13 (Estimated); Status verified 2009-05

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal reflux disease; Mosapride; Lansoprazole
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — mosapride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): lansoprazole plus mosapride for the first month, and followed by lansoprazole plus placebo for the second month
  Interventions: Drug: mosapride for the first month and placebo for the 2nd month
- 2 (Active Comparator): lansoprazole plus placebo for the first month, and lansoprazole plus mosapride for the second month
  Interventions: Drug: placebo for the first and mosapride for the second month

INTERVENTIONS:
Drug: mosapride for the first month and placebo for the 2nd month — lansoprazole 30 mg once per day for 2 months mosapride 5 mg thrice per day, for the first month placebo thrice per day, for the second month
  Arms: 1
Drug: placebo for the first and mosapride for the second month — lansoprazole 30 mg once per day for 2 months placebo thrice per day, for the first month mosapride 5 mg thrice per day, for the second month
  Arms: 2

SUMMARY:
Gastroesophageal reflux disease (GERD) is a very common disease in the Western World. In Taiwan, this disease is increasing gradually because the investigators' eating style is closing to Western world.

Proton pump is the main drug for patients with GERD in the past two decades. Prokinetic agent is an important adjuvant to the therapy of GERD. This study aims to evaluate the role of prokinetic agent in the management of GERD.

DETAILED DESCRIPTION:
This is a randomized, double-blind, cross-over study. FSSG is obtained at the beginning, one month and two months of the study.

This study plans to enroll 100 patients with symptoms of GERD (acid regurgitation, belching, dysphagia). After receiving endoscopic examination, a frequent scale for the symptoms of gastroesophageal reflux disease (FSSG) is obtained from these patients. Fifty patients receive lansoprazole 30 mg once plus mosapride 5 mg tid daily in the first month; and lansoprazole 30 mg once plus placebo tid daily in the second month. Another fifty patients receive lansoprazole 30 mg once plus placebo tid daily in the first month; and lansoprazole 30 mg once plus mosapride 5 mg tid daily in the second month.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 90 years old
* Outpatients
* Characteristic GERD symptoms: acid regurgitation, heart burn, or belching
* Erosive esophagitis on upper digestive endoscopy, based on Los Angeles classification

Exclusion Criteria:

* History of allergy to lansoprazole or mosapride
* Pregnant or lactating women
* Uremia
* Decompensated liver disease
* Age under 18 and over 90 years-old
* Lack of informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2008-06; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Symptom improvement evaluated by frequent scale for the symptoms of gastroesophageal reflux disease (FSSG) | before enrollment, one month after treatment, two months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hwai-Jeng Lin, M.D., Principal Investigator — Lotung Poh-Ai Hospital
Locations (1):
- Lotung Poh-Ai Hospital, Lotung Town, Ilan County, Taiwan